CLINICAL TRIAL: NCT00921050
Title: Randomized Double Blind Levothyroxine vs Placebo, Mind (NEUROPSI) Improvement in Elderly With Persistent TSH 4-10 mUI/L
Brief Title: Subclinical Hypothyroidism and Mind in the Elderly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Lilia Csrdenas-Ibarra, MD, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EN_LC_P136
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Subclinical Hypothyroidism
Keywords: subclinical hypothyroidism; elderly; mild cognitive impairment; neuropsychological test; NEUROPSI
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Thyroxine; Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levothyroxine (Experimental): Half of participants randomly assigned, take a pill daily, bimonthly thyroid test
  Interventions: Drug: levothyroxine sodium
- Placebo (Placebo Comparator): Half of participants randomly assigned, take a pill daily, bimonthly thyroid test
  Interventions: Drug: excipient without levothyroxine (placebo)

INTERVENTIONS:
Drug: levothyroxine sodium — Daily intake (fasting) levothyroxine bimonthly adjusted; to keep TSH between 0.5 to 2.5 mUI/L range. Start with 12.5mcg an investigator other than the caregiver will review the TSH measurements to adjust levothyroxine dose that will contain the coded bottle with the pils given to patient.
  Other Names: eutirox (Merck); synthroid
  Arms: Levothyroxine
Drug: excipient without levothyroxine (placebo) — Daily intake (fasting) a pill. bimonthly adjusted; an investigator other than the caregiver will review the TSH measurements and pretend to adjust dose contained in the coded bottle with the pills given to patient.
  Other Names: sugar pills
  Arms: Placebo

SUMMARY:
Some recommendations of expert consensus on subclinical hypothyroidism (SH) are controversial in those areas with not enough information to reach a conclusion, such as not recommending treatment with thyrotrophic hormone of 4-10 mUI/L and free thyroxin in normal range. The body changes or symptoms at this stage are often mistaken as aging. There are studies showing significant changes in heart (slow rate, lower ejection fraction, diastolic dysfunction); hypercholesterolemia, dysfunction cognitive abilities (memory attention…).

The prevalence of SH increases with age, reaching 14% over 65 years old. This age group increase as the population ages highlights the need for evidence to improve recommendations for the elderly.

NEUROPSI is a validated neuropsychological test sensible for mild cognitive alterations. It can be applied to individuals with little schooling.

This study aims to determine positive change in cognitive abilities (NEUROPSI), ejection fraction, and body percent of lean and adipose tissue without adverse effects, placebo versus thyroxin supplement to keep thyroid-stimulating hormone (TSH) between 0.5-2.5 mUI/L in elderly with TSH 4-10 mIU/L.

DETAILED DESCRIPTION:
Screening, subjects > 59 y/o with out exclusion criteria to identify HS, started in October 15, 2008. Due to difficulties getting the placebo for the assay, by January halted the screening. At the end of May we got the donation from Merck pharmaceuticals.

The protocol original dates changed as follows:

* Restart screening June 20 to end in August 2009;
* Enrolling start at the end of June (the already identified);
* End enrolling October 2009;
* Follow up will end in May 2010.

Note: 150 of the screened subjects will be from randomly selected homes at Fomerrey 19 to allow prevalence estimation.

* Enroling ended until june 2010
* Follow up stil ungoing final measures will be done at the end of 2011

ELIGIBILITY:
Inclusion Criteria:

* TSH between 4 and 10 mUI/L inclusive

Exclusion Criteria:

* Known and treatment of thyroideal disease
* Arrythmia
* Anticoagulant treatment
* Dementia
* Disease leading to dementia (acv, LIVER....)

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in cognitive ability measured by NEUROPSI increase of 10 points | baseline and after 6 months of treatment
ejection fraction, left ventricular diastolic capacity | baseline, after six months of treatment
Lipid profile and body composition by DEXA | baseline, after six months of treatment

SECONDARY OUTCOMES:
clinical assessment v.g. significant changes in cardiac frequency and rhythm (if needed able to take EKG to confirm) | bimonthly
Free tiroxina and TSH (assessed by investigator other than treatment physician) | bimonthly
Changes in EKG | baseline, at six months, or as needed

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Cardenas-Ibarra, M.D., Principal Investigator — Endocrinology, University Hospital, Universidad Autonoma de Nuevo Leon; Jesus Z Villarreal-Perez, M.D., Study Chair — Endocrinology, University Hospital, Universidad Autonoma de Nuevo Leon
Locations (2):
- Mexico (2):
  - Endocrinology, Outpatient Hospital Clinic, Monterrey, Nuevo León
  - Community Health Center (Fomerrey 19), Monterrey, Nuevo León